CLINICAL TRIAL: NCT03312348
Title: High Resolution Infrared Thermographic Imaging as a Diagnostic Aid for Acute Undifferentiated Limp in Children.
Brief Title: High Resolution IR Imaging for Diagnosis in the Acute Limping Child - ThermLimp
Acronym: Thermlimp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCH-13-067C
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Results first posted 2019-04-24 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Limping
MeSH Terms: conditions — Intermittent Claudication

ARMS (1):
- Infrared Imaging undertaken (Experimental): Infrared imaging of Region Of Interest in study participants
  Interventions: Device: Infrared imaging

INTERVENTIONS:
Device: Infrared imaging — Infrared image image acquisition of study participants

SUMMARY:
A variety of different diseases may cause a limp in a child, and in younger children it is particularly challenging to isolate the area affected. Children of this age group are unable to identify a specific region of pain, so clinical examination and parental interpretation is the only method of localising the area of discomfort. Potential problems that may affect children include inflammation, fractures, infection, juvenile arthritis or movement in the growth plate in the hip, among other diseases. Aside from an obvious source of injury, it is challenging for a clinician to distinguish between these different potential causes or the area of the problem without repeated visits, non-specific blood tests and the use of x-ray imaging: a form of radiation that carries with it a small risk of carcinogenic effect. Once a region of the lower limb is identified, an x-ray image of the affected area is often taken; however, it is not possible to image the entire leg, so the importance of the initial examination by a clinician is evident. The aim of this research project is to assess the potential of high resolution infrared (IR) imaging technology in the identification of a focus for the cause of a limping child. The IR camera used for imaging is able to observe an entire limb, so the need to localise an area for imaging would be removed. In addition, if successful, infrared imaging could reduce the number of children exposed to x-ray radiation unnecessarily, whilst stream-lining medical practice by reducing the time to make a diagnosis along with unnecessary visits and tests. The investigators aim to explore whether non-invasive IR thermographic camera imaging assists with the clinical diagnosis in children presenting with an acute limp. This study represents a pilot evaluation as a test of concept.

ELIGIBILITY:
Inclusion Criteria:

* Children age 9 months -16 years old who attend the Emergency Department (ED) of the Sheffield Children's Hospital for an acute (less than 48 hours) limp. Inclusion is subject to both the patient and carer having read (or being read to in very young children) the information sheets and both the patient and carer consenting to participate.

Exclusion Criteria:

* Children with multiple injuries (e.g. those involved in serious car accidents), or those who have difficulty understanding the nature of the study (e.g. non-native English speakers, those with disabilities impairing their understanding of the study etc.) will be excluded. Patients/carers in whom consent has not been obtained or refused will also be excluded.

Children who attend the ED with safeguarding concerns or in whom child protection suspicions arise during the consultation will be excluded. These children have a separate assessment process which would be significantly different to the study cohort.

Ages: 9 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06-30 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infrared Imaging Undertaken
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infrared Imaging Undertaken
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.2 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Which Thermal Imaging Technique Correctly Identified Area of Focus for a Limping Child
Description: Number of Participants for Which Thermal Imaging Technique Correctly Identified Area of Focus for a Limping Child - 25
Time Frame: 10 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Infrared Imaging Undertaken
Number analyzed (Participants) | 30
Participants | 30

ADVERSE EVENTS:
Time Frame: Adverse event data was requested for 6 months after recruitment.
Arm/Group | Infrared Imaging Undertaken
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes